CLINICAL TRIAL: NCT05905523
Title: Testing of Online Version of QAPS
Status: Recruiting | Type: Observational
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Other Study IDs: HM20026549
Record Dates: First submitted 2023-06-07; First posted 2023-06-15 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Child Development

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- 3 year old participants: In this study, your child will be asked to do the following things:
  1. Play a drawing game on a tablet
  2. Copy shapes using a pencil in a paper booklet
  3. Write some letters and cut paper with scissors You will complete surveys and answer questions about your child's development
  Interventions: Other: Assessing prewriting skills in children
- 4 year old participants: In this study, your child will be asked to do the following things:
  1. Play a drawing game on a tablet
  2. Copy shapes using a pencil in a paper booklet
  3. Write some letters and cut paper with scissors You will complete surveys and answer questions about your child's development
  Interventions: Other: Assessing prewriting skills in children
- 5 year old participants: In this study, your child will be asked to do the following things:
  1. Play a drawing game on a tablet
  2. Copy shapes using a pencil in a paper booklet
  3. Write some letters and cut paper with scissors You will complete surveys and answer questions about your child's development
  Interventions: Other: Assessing prewriting skills in children
- 6 year old participants: In this study, your child will be asked to do the following things:
  1. Play a drawing game on a tablet
  2. Copy shapes using a pencil in a paper booklet
  3. Write some letters and cut paper with scissors You will complete surveys and answer questions about your child's development
  Interventions: Other: Assessing prewriting skills in children
- 7 year old participants: In this study, your child will be asked to do the following things:
  1. Play a drawing game on a tablet
  2. Copy shapes using a pencil in a paper booklet
  3. Write some letters and cut paper with scissors You will complete surveys and answer questions about your child's development
  Interventions: Other: Assessing prewriting skills in children

INTERVENTIONS:
Other: Assessing prewriting skills in children — In this study, your child will be asked to do the following things:
  1. Play a drawing game on a tablet
  2. Copy shapes using a pencil in a paper booklet
  3. Write some letters and cut paper with scissors You will complete surveys and answer questions about your child's development

SUMMARY:
Early evaluation of prewriting skills is important, as prewriting skills set the stage for later learning of the fine motor and visual motor skills needed for writing. Evaluation of prewriting skills allows for the identification of those children who struggle with these tasks so that early intervention might address these foundational skills before academic demands become more challenging. However, current prewriting skill assessments are limited to pencil-and-paper assessments that require an evaluator to score the drawn shapes. Manual scoring is time consuming, can be subjective, and limit the ability to capture subtle changes in performance.

We have developed an assessment on a tablet to assess prewriting skills in children. The preliminary testing of the assessment is published in a paper (https://pubmed.ncbi.nlm.nih.gov/35417278/). We are now working on developing an online version of the assessment that will allow offsite data collection and will automate the analysis on the website so that the results can be automatically generated for the clinician or educator who wants to use this with the children they work with.

ELIGIBILITY:
Inclusion Criteria:

* Children between 3 to 7 years old

Exclusion Criteria:

* Children unable to follow directions to attempt copying shapes.

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children between 3 to 7 years old
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-10-03 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Online QAPS | 5-10 minutes
  Children will be asked to draw shapes on a touch-screen tablet, where the top half of the screen will show the shapes that they needed to draw, and the bottom of half of the screen will show a space for them to copy the shape. There are 10 shapes for the children to copy. This assessment takes 5-10 minutes to complete.
Beery VMI | 5-10 minutes
  This is a pencil-paper visual motor assessment where children are asked to copy the shapes of increasing difficulty. There are 24 shapes in this assessment and the assessment is continued until the child cannot copy 3 consecutive shapes. This assessment takes 5-10 minutes to complete.
Functional hand tasks | 5-10 minutes
  We will have the children demonstrate their handwriting and scissors skills. The tasks that the children as asked to complete is listed in the attached documents. This assessment takes 5-10 minutes to complete.
Demographics survey | 5 minutes
  This is a 12 question survey that ask about the child's age, grade level, sex, race, caregiver education level, household income, state of residency, etc. This survey should take about 5 minutes to complete.
Emotionality Assessment | 5 minutes
  This is a 5 question survey that asks the caregiver to rate the child's ability to regulate emotions. This survey should take about 5 minutes to complete.
Strengths & difficulties Questionnaire Inattention/Hyperactivity subscale | 5 minutes
  This is a 5 question survey that asks the caregiver to rate the child's attentional behavior. This survey should take about 5 minutes to complete.
Ego Resiliency Scale | 5 minutes
  This is a 11 question survey that asks the caregiver to rate the child's ability to adapt to change. This survey should take about 5 minutes to complete.

CONTACTS AND LOCATIONS:
Overall Officials: Virginia Chu, PhD, OTR/L, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonweath University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No